CLINICAL TRIAL: NCT00762385
Title: Clinical Comparison of Two Silicone-Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Foresight Regulatory Strategies, Inc. (Industry); Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0713
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- galyfilcon A/comfilcon A (Active Comparator): galyfilcon A first, comfilcon A second
  Interventions: Device: galyfilcon A; Device: comfilcon A
- comfilcon A/galyfilcon A (Active Comparator): comfilcon A first, galyfilcon A second
  Interventions: Device: galyfilcon A; Device: comfilcon A

INTERVENTIONS:
Device: galyfilcon A — galyfilcon A
Device: comfilcon A — comfilcon A

SUMMARY:
The objective of this study is to evaluate the clinical performance of two silicone-hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 and less than or equal to 39 years of age and have a need for vision correction in both eyes.
* The subject must require a lens power between -1.00 to -6.00D and have no more than 1.00D of corneal cylinder.
* The subject, based on his/her knowledge, must be in good general health.
* The subject must be able and willing to adhere to the instructions set forth in this protocol and complete all specified evaluations.
* Subject must be a current adapted daily wearer of soft contact lenses with at least 6 months of CL wear.
* Subject must agree to wear their contact lenses in both eyes on a daily wear schedule for at least 8 hours per day every day during the study.
* Subject must be willing and able to use only the care systems and lubricating drops provided for the study during the 4 week period.
* The subject must read, indicate understanding of and sign the Informed Consent Form.

Exclusion Criteria:

* The subject is a rigid gas permeable (RGP) or daily disposable lens wearer.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids or associated structures.
* The presence of ocular or systemic disease or need for medication which might interfere with contact lens wear or which would cause the lenses to be removed more than twice a day. (i.e., Sjogren's syndrome, type II diabetes, etc.)
* Slit lamp findings that would contraindicate contact lens wear such as:

  * pathological dry eye or associated findings
  * pterygium or corneal scars within the visual axis
  * neovascularization equal to or greater than 1mm in from the limbus
  * history of giant papillary conjunctivitis (GPC) worse than grade 2
  * anterior uveitis or iritis (past or present)
  * seborrhoeic eczema
  * seborrhoeic conjunctivitis
* A history of recurrent erosions, corneal infiltrates, corneal ulcer or fungal infections.
* A known history of corneal hypoesthesia (reduced corneal sensitivity).
* Contact lens snellen visual acuities (VA) worse than 20/30.
* Aphakia, keratoconus or a highly irregular cornea.
* Current pregnancy or lactation (to the best of the subject's knowledge)
* Any active participation in another clinical study at any time during this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Galyfilcon A / Comfilcon A: galyfilcon A contact lenses first period, comfilcon a contact lenses second period
- Comfilcon A / Galyfilcon A: comfilcon A contact lenses first period, galyfilcon A contact lenses second period
Period: First Intervention
Arm/Group | Galyfilcon A / Comfilcon A | Comfilcon A / Galyfilcon A
Started | 51 | 46
Completed | 49 | 42
Not Completed | 2 | 4
Not completed — Lens Issue | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Ineligible | 1 | 0
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention
Arm/Group | Galyfilcon A / Comfilcon A | Comfilcon A / Galyfilcon A
Started | 49 | 42
Completed | 46 | 39
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Completed Population: Includes subjects randomized to galyfilcon A/comfilcon A and comfilcon A/galyfilcon A and that completed the study.
Arm/Group | Completed Population
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Lens Comfort
Description: >0 = comfortable, <0 = uncomfortable; a weighted combined score calculated from individual comfort-related questions was used to derive comfort outcomes.
Time Frame: 1-week, 2- weeks
Population: Only participants who completed the study per protocol (n=78)
Measure: Least Squares Mean (Standard Error); unit: combined score
Groups:
- Galyfilcon A: galyfilcon A administered in either the first intervention period or the second intervention period.
- Comfilcon A: comfilcon A administered in either the first intervention period or second intervention period.
Arm/Group | Galyfilcon A | Comfilcon A
Number analyzed (Participants) | 78 | 78
combined score | 0.1452 (0.1097) | 0.1135 (0.1112)
Statistical Analysis 1: Comparison: Galyfilcon A vs Comfilcon A; Results is overall lens effect with time as a covariate; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.03164, 98.3% CI [-0.2346 to 0.03164], Standard Error of Mean 0.1247 — Mean difference is galyfilcon A minus comfilcon A

2. Secondary Outcome: Overall Corneal Staining
Description: Measured for 5 zones of the cornea (superior, nasal, central, inferior, temporal)on a 0 to 3 grade scale (NEI 0-3 scale). Grade 0 = Normal/ grade 1 = mild, superficial stippling/ grade 2 = moderate, punctate staining including superficial abrasion of the cornea/ grade 3 = severe, abrasion or corneal erosion, deep corneal abrasion or recurrent erosion.
Time Frame: 2 weeks
Population: Only the participants who completed the study per protocol (n=78)
Measure: Least Squares Mean (Standard Error); unit: combined score
Arm/Group | Galyfilcon A | Comfilcon A
Number analyzed (Participants) | 78 | 78
combined score | 0.07582 (0.02192) | 0.07026 (0.02192)
Statistical Analysis 1: Comparison: Galyfilcon A vs Comfilcon A; Results is overall lens effect with time as a covariate; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.005560, 98.3% CI [-0.04297 to 0.005560], Standard Error of Mean 0.02287 — Mean difference is galyfilcon A minus comfilcon A

3. Primary Outcome: Comfort Symptoms
Description: A weighted combined score calculated from individual comfort-related questions was used to derive comfort outcomes. >0 = comfortable, <0 = uncomfortable
Time Frame: 1-week, 2-weeks
Population: Only participants who completed the study per protocol (n=78)
Measure: Least Squares Mean (Standard Error); unit: score
Groups:
- Comfilcon A: comfilcon A administered in either the first intervention period or the second intervention period.
Arm/Group | Galyfilcon A | Comfilcon A
Number analyzed (Participants) | 78 | 78
score | 0.2440 (0.1262) | -0.02862 (0.1275)
Statistical Analysis 1: Comparison: Galyfilcon A vs Comfilcon A; Results is overall lens effect with time as a covariate; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.2726, 98.3% CI [0.04553 to 0.2726], Standard Error of Mean 0.1064 — Mean difference is galyfilcon A minus comfilcon A

ADVERSE EVENTS:
Arm/Group | Galyfilcon A / Comfilcon A | Comfilcon A / Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/46
Other Adverse Events (participants affected / at risk) | 0/51 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.